CLINICAL TRIAL: NCT04216797
Title: Rectal Versus Oral Diazepam Administration in the Treatment of Levator Ani Syndrome in Participants Who Have Not Responded to Physical Therapy Treatment: A Prospective Randomized Study
Brief Title: Rectal Versus Oral Diazepam Administration in the Treatment of Levator Ani Syndrome
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment was initially suspended due to COVID pandemic. As the number of cases subsided, enrollment was reopened but never regained momentum. PI has left the site.
Sponsor: Swedish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY2019000291
Record Dates: First submitted 2019-12-23; First posted 2020-01-03 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-02

CONDITIONS: Levator Ani Syndrome
MeSH Terms: conditions — Levator syndrome | interventions — Diazepam

STUDY DESIGN:
Intervention Model Description: All participants will initially receive 6 weeks of pelvic floor PT. After these six weeks, qualifying participants will be randomized to one of two arms: rectal or oral diazepam administration. Participants will be dispensed 30, 10 mg diazepam tablets to take daily (oral or rectal) for 4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Administration (Active Comparator): 10 mg diazepam tablets to be taken orally once daily for 4 weeks.
  Interventions: Drug: Diazepam Tablets
- Rectal Administration (Active Comparator): 10 mg diazepam tablets to be taken rectally once daily for 4 weeks.
  Interventions: Drug: Diazepam Tablets

INTERVENTIONS:
Drug: Diazepam Tablets — Participants will be randomly assigned to either an oral or rectal administration of once daily 10 mg diazepam tablets for four weeks.

SUMMARY:
This research involves collecting data about levator ani syndrome (LAS) associated rectal pain and a comparison of diazepam treatment administration routes. The goal of this research is to see if an alternative route of diazepam administration provides sufficient control of LAS discomfort and low sleep quality while minimizing systemic effects of diazepam (drowsiness).

DETAILED DESCRIPTION:
Levator ani syndrome (LAS) is described as a dull, aching pain of a patient's pelvic floor musculature. There is no known cause for the syndrome, yet pelvic floor muscle spasm and increased anal resting pressures have been hypothesized to result in the syndrome. LAS is commonly seen in patients with constipation, specifically outlet dysfunction constipation. Treatment for the syndrome involves a combination of bowel management, medications, and pelvic floor physical therapy (PT). Pelvic floor PT uses a variety of methods to help patients with LAS, including biofeedback and massage. The literature and the investigators experience shows that these pelvic floor PT approaches do not resolve all LAS symptoms.

Diazepam (Valium®) is used to treat levator ani syndrome in conjunction with other treatments to help relax the pelvic floor muscle group (levator ani). Diazepam has U.S. Food and Drug Administration (FDA) approval for use as a muscle relaxant. Investigators at Swedish Colon & Rectal Clinic are using diazepam intervention as a means for patients to gain relief from pain.

The work proposed aims to provide the first prospective, randomized, comparative study of the efficacy between administering diazepam rectally and administering the medication orally after pelvic floor PT treatment. Currently, other ways of administering diazepam have not been studied in the setting of the LAS condition. The Investigators performed a retrospective chart review last year and found some promising results for the efficacy of rectal and oral routes of diazepam for LAS. The Investigators want to determine if the route of administering diazepam as an adjunct to pelvic floor PT influences rectal pain relief for LAS patients.

Primary Objective: Compare the pain scores of participants with LAS after administering diazepam rectally or orally following six weeks of physical therapy.

Secondary Objectives:

1. Measure and compare the drowsiness levels of participants using rectal diazepam or oral diazepam. 2. Measure and compare the sleep quality of participants using rectal diazepam or oral diazepam.

All participants with the LAS diagnosis will initially receive 6 weeks of pelvic floor PT. After these six weeks, participants without effective pain relief will be randomized to one of two arms: rectal or oral diazepam administration. Participants will be dispensed 30 10 mg diazepam tablets to take daily (oral or rectal) for 4 weeks. Participants will be asked to complete 3 electronic questionnaires (VAS pain scale, Likert drowsiness scale, and Pittsburg Sleep Quality Index) each week while on the 10 week trial. Investigators plan to enroll 100 participants over approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of LAS according to the Rome IV criteria with:

   1. Chronic or recurrent rectal pain or aching
   2. Episodes lasting 30 minutes or longer
   3. Tenderness during traction on the puborectalis
   4. Exclusion of other causes of rectal pain
2. Patients who agree to undergo pelvic floor PT for six weeks prior to starting the medication treatment.
3. Women ≥ 18 years of age. Women of childbearing potential must undergo urine pregnancy testing prior to using the treatment medication.
4. Men ≥ 18 years of age.

Exclusion Criteria:

1. Participants who have had pelvic floor surgery or with recent conditions in which rectal suppositories are contraindicated.
2. Non-English speaking participants.
3. Women who are pregnant or breastfeeding.
4. Participants who are cognitively impaired, illiterate, or have a condition in which they are unable to consent for themselves.
5. Prisoners.
6. Participants allergic to benzodiazepines or have a sensitivity/intolerance to benzodiazepines.
7. Participants to which benzodiazepines are contraindicated or are on medications that interact with benzodiazepines.
8. Participants with current or history of Diagnostic and Statistical Manual of Mental Disorders (DSM-V) substance use disorder or Participants with a history of evidence of severe illness or any other conditions that would affect absorption or make the patient unsuitable for the study in the opinion of the investigator.
9. Participants already receiving medications in the benzodiazepine class within 2 weeks of screening visit for any reasons will be excluded based on increased risk for medication tolerance.
10. Participants who have undergone pelvic floor PT within 2 weeks of screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
Effectiveness of rectal administration versus oral administration in LAS pain management: Visual Analog Scale (VAS) | 10 weeks
  Participants will complete weekly electronic Visual Analog Scale (VAS) for pain for 6 weeks while on Physical Therapy only, followed by 4 weeks while taking diazepam (orally or rectally). Participants will be asked to select a number on a scale of 1 to 10, where 1 equals no pain and 10 equals worst pain.

SECONDARY OUTCOMES:
Participant drowsiness while taking diazepam rectally versus orally | 10 weeks
  Participants will complete weekly electronic Likert drowsiness scale for 6 weeks while on Physical Therapy only, followed by 4 weeks while taking diazepam (orally or rectally). Participants will be asked to select a number on a scale of 1 to 5, where 1 equals much less drowsiness than usual and 10 equals much more drowsiness than usual.
Participant sleep quality while taking diazepam rectally versus orally: Pittsburg Sleep Quality Index | 10 weeks
  Participants will complete weekly electronic Pittsburg Sleep Quality Index for 6 weeks while on Physical Therapy only, followed by 4 weeks while taking diazepam (orally or rectally).
  The Pittsburg Sleep Quality Index measures overall sleep quality, evaluating seven categories of sleep: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
  The seven individual categories are weighted on a 0-3 interval scale. The global Pittsburg Sleep Quality Index score is then calculated by adding the seven individual category scores, which then provides a total score ranging from 0 to 21, where lower scores represent a healthier sleep quality.
Study Medication Adherence | 4 weeks
  Participants will be instructed to take diazepam (orally or rectally) daily for 4 weeks. Participants will bring in their pill bottles so that the study staff can manually count their pills to check for adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia A Lynn, Principal Investigator — Swedish Medical Center
Locations (1):
- Swedish Medical Center Colon Rectal Clinic, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No